CLINICAL TRIAL: NCT06231667
Title: The Effect of Health Literacy Education Given in Early Adolescence on Adolescents' Health Literacy
Brief Title: The Effect of Health Literacy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Prof. Dr., Dean of the Faculty of Nursing, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/07.03.2022
Record Dates: First submitted 2024-01-18; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Health Literacy Level
Keywords: health literacy; education; adolescent
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): The health literacy training was implemented in a total of 4 sessions, each session lasting 30 minutes, with an interval of one week. Various teaching methods and techniques were used in the trainings.
  Interventions: Other: Education
- Control (No Intervention)

INTERVENTIONS:
Other: Education — four training sessions were applied to the intervention group
  Arms: Education

SUMMARY:
The study was conducted with a parallel group randomized controlled experimental design to evaluate the effect of health literacy education given in early adolescence on the health literacy of adolescents. The population of the study consisted of 6th and 7th grade (12-13 years old) students studying in a secondary school in Ankara. Power analysis was used to determine the sample size. A total of 80 adolescents who met the inclusion criteria were included in the sample.

ELIGIBILITY:
Inclusion Criteria:

* Consent by the student's family
* Volunteering to participate in the research
* Having a low level of health literacy

Exclusion Criteria:

* Read and write Turkish
* Have a moderate or high level of health literacy
* Physical/mental disability or illness

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Health Literacy Level (School Age Children Health Literacy Scale) | before the implementation
  Health literacy level was evaluated in three groups: low health literacy (10-25 points), moderate health literacy (26-35 points) and (36-40) points: high health literacy (36-40 points). Intervention and control groups were selected among the students with low health literacy levels.
Health Literacy Level (School Age Children Health Literacy Scale) | one month after the education
  Health literacy level was evaluated in three groups: low health literacy (10-25 points), moderate health literacy (26-35 points) and (36-40) points: high health literacy (36-40 points). Intervention and control groups were selected among the students with low health literacy levels.
Health Literacy Level (School Age Children Health Literacy Scale) | three month after the education
  Health literacy level was evaluated in three groups: low health literacy (10-25 points), moderate health literacy (26-35 points) and (36-40) points: high health literacy (36-40 points). Intervention and control groups were selected among the students with low health literacy levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)